CLINICAL TRIAL: NCT03417778
Title: A Phase 1 Open-Label Study to Evaluate the Pharmacokinetics of Filgotinib in Subjects With Impaired Hepatic Function
Brief Title: Study to Evaluate the Pharmacokinetics of Filgotinib in Participants With Impaired Hepatic Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Collaborators: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GS-US-417-4048; 2017-000156-25 (EudraCT Number)
Record Dates: First submitted 2018-01-25; First posted 2018-01-31 (Actual); Results first posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2020-12

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — GLPG0634

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Moderate Hepatic Impairment (Experimental): Participants with moderate hepatic impairment and matched healthy controls will receive a single dose of filgotinib on Day 1.
  Interventions: Drug: Filgotinib
- Severe Hepatic Impairment (Experimental): Participants with severe hepatic impairment and matched healthy controls will receive a single dose of filgotinib on Day 1.
  Interventions: Drug: Filgotinib
- Mild Hepatic Impairment (Experimental): Participants with mild hepatic impairment and matched healthy controls will receive a single dose of filgotinib on Day 1.
  Interventions: Drug: Filgotinib

INTERVENTIONS:
Drug: Filgotinib — 100 mg tablet administered orally
  Other Names: GS-6034; GLPG0634

SUMMARY:
The primary objective of this study is to evaluate the pharmacokinetics (PK) of filgotinib and its metabolite, GS-829845, in participants with varying degrees of impaired hepatic function relative to matched, healthy controls.

ELIGIBILITY:
Key Inclusion Criteria:

* Eligible individuals will be male and nonpregnant, nonlactating females, aged 18 to 70 years (inclusive), body mass index (BMI) between 18 and 36 kg/m^2 (inclusive), with either impaired hepatic function or normal hepatic function.
* Individuals will be current nonsmokers (no use of tobacco, nicotine-containing, or tetrahydrocannabinol [THC]-containing products within the last 14 days).
* Individuals with hepatic impairment will be categorized by the Child-Pugh-Turcotte (CPT) classification system indicating hepatic impairment as follows:

  * Class A (mild): CPT score 5-6
  * Class B (moderate): CPT score 7-9
  * Class C (severe): CPT score 10-15
* Hepatic impairment must have been stable during the 3 months (90 days) prior to study drug. Each individual in the control group will be matched to a individual with impaired hepatic function by age (± 10 years), gender, and body mass index (± 15%).

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-04-03 (Actual); Primary Completion 2018-08-09 (Actual); Study Completion 2018-08-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (4):
- United States (2):
  - Clinical Pharmacology of Miami, Miami, Florida
  - American Research Corporation at the Texas Liver Institute, San Antonio, Texas
- APEX GmbH, Munich, Germany
- Auckland Clinical Studies Ltd., Grafton, Auckland, New Zealand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Anderson K, Zheng H, Medzihradsky O, et al. THU0117 PHARMACOKINETICS AND SHORT-TERM SAFETY OF FILGOTINIB, A SELECTIVE JANUS KINASE 1 INHIBITOR, IN SUBJECTS WITH MODERATE HEPATIC IMPAIRMENT. Annals of the Rheumatic Diseases. 2019;78:331.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Germany, New Zealand, and United States. The first participant was screened on 03 April 2018. The last study visit occurred on 09 August 2018.
Pre-assignment Details: 38 participants were screened. Per protocol, participants in adaptive Cohort 2 (severe hepatic impairment) and Cohort 3 (mild hepatic impairment) were not enrolled following review of safety and pharmacokinetic (PK) data from participants in Cohort 1 (moderate hepatic impairment).
Groups:
- Moderate Hepatic Impairment: Participants with moderate hepatic impairment received a single dose of filgotinib 100 mg administered orally on Day 1, in a fasted state.
- Healthy Control: Matched healthy control participants received a single dose of filgotinib 100 mg administered orally on Day 1, in a fasted state.
Period: Overall Study
Arm/Group | Moderate Hepatic Impairment | Healthy Control
Started | 10 | 10
Completed | 10 | 10
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set included all enrolled participants who received at least 1 dose of study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Moderate Hepatic Impairment | Healthy Control | Total
Number analyzed (Participants) | 10 | 10 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 61 (6.9) | 62 (5.3) | 61 (6.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 14
  Male | 3 | 3 | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 5 | 10
  Not Hispanic or Latino | 5 | 5 | 10
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 10 | 10 | 20
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  New Zealand | 2 | 2 | 4
  United States | 6 | 6 | 12
  Germany | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetic (PK) Parameter: AUClast of Filgotinib
Description: AUClast is defined as the concentration of drug from time zero to the last observable concentration.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36, 48, 72, 96, and 120 hours postdose on Day 1
Population: The PK Analysis Set included all enrolled participants who received at least 1 dose of filgotinib and had at least 1 nonmissing postdose concentration value of filgotinib or its primary metabolite GS-829845 reported by the PK laboratory.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Moderate Hepatic Impairment | Healthy Control
Number analyzed (Participants) | 10 | 10
h*ng/mL | 2389.3 (530.85) | 1981.9 (995.78)
Statistical Analysis 1: Comparison: Moderate Hepatic Impairment vs Healthy Control; An analysis of variance (ANOVA) model was fitted to the natural logarithmic transformed values of the AUClast. Two-sided 90% confidence intervals (CI) were calculated for the geometric least-squares mean (GLSM) ratio of AUClast between hepatic impairment group versus the matched control (normal hepatic function) group; Test type: Other — If the upper bound of the 2-sided 90% CIs of the GLSM ratio for AUClast of filgotinib falls within the [50%, 200%] bound, the null hypothesis that participants with hepatic impairment exhibit AUClast change of at least 2-fold for filgotinib compared with participants with normal liver function will be rejected; GLSM Ratio = 161.14, 90% CI 2-sided [80.77 to 321.48]

2. Primary Outcome: PK Parameter: AUClast of GS-829845
Description: AUClast is defined as the concentration of drug from time zero to the last observable concentration. GS-829845 is the primary metabolite of filgotinib.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36, 48, 72, 96, and 120 hours postdose on Day 1
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Moderate Hepatic Impairment | Healthy Control
Number analyzed (Participants) | 10 | 10
h*ng/mL | 32466.8 (10898.85) | 31412.6 (13758.34)
Statistical Analysis 1: Comparison: Moderate Hepatic Impairment vs Healthy Control; An ANOVA model was fitted to the natural logarithmic transformed values of the AUClast. Two-sided 90% CI were calculated for the GLSM ratio of AUClast between hepatic impairment group versus the matched control (normal hepatic function) group; Test type: Other — If the upper bound of the 2-sided 90% CIs of the GLSM ratio for AUClast of GS-829845 falls within the [50%, 200%] bound, the null hypothesis that participants with hepatic impairment exhibit AUClast change of at least 2-fold for GS-829845 compared with participants with normal liver function will be rejected; GLSM Ratio = 122.08, 90% CI 2-sided [69.67 to 213.89]

3. Primary Outcome: PK Parameter: AUCinf of Filgotinib
Description: AUCinf is defined as the concentration of drug extrapolated to infinite time.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36, 48, 72, 96, and 120 hours postdose on Day 1
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Moderate Hepatic Impairment | Healthy Control
Number analyzed (Participants) | 10 | 10
h*ng/mL | 2417.0 (533.74) | 1995.9 (997.88)
Statistical Analysis 1: Comparison: Moderate Hepatic Impairment vs Healthy Control; An ANOVA model was fitted to the natural logarithmic transformed values of the AUCinf. Two-sided 90% CI were calculated for the GLSM ratio of AUCinf between hepatic impairment group versus the matched control (normal hepatic function) group; Test type: Other — If the upper bound of the 2-sided 90% CIs of the GLSM ratio for AUCinf of filgotinib falls within the [50%, 200%] bound, the null hypothesis that participants with hepatic impairment exhibit AUCinf change of at least 2-fold for filgotinib compared with participants with normal liver function will be rejected; GLSM Ratio = 159.15, 90% CI 2-sided [82.22 to 308.06]

4. Primary Outcome: PK Parameter: AUCinf of GS-829845
Description: AUCinf is defined as the concentration of drug extrapolated to infinite time. GS-829845 is the primary metabolite of filgotinib.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36, 48, 72, 96, and 120 hours postdose on Day 1
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: h*ng/mL
Arm/Group | Moderate Hepatic Impairment | Healthy Control
Number analyzed (Participants) | 10 | 10
h*ng/mL | 33296.5 (11568.33) | 32060.0 (14329.57)
Statistical Analysis 1: Comparison: Moderate Hepatic Impairment vs Healthy Control; [analysis description as in outcome 3, analysis 1]; Test type: Other — If the upper bound of the 2-sided 90% CIs of the GLSM ratio for AUCinf of GS-829845 falls within the [50%, 200%] bound, the null hypothesis that participants with hepatic impairment exhibit AUCinf change of at least 2-fold for GS-829845 compared with participants with normal liver function will be rejected; GLSM Ratio = 122.32, 90% CI 2-sided [69.90 to 214.07]

5. Primary Outcome: PK Parameter: Cmax of Filgotinib
Description: Cmax is defined as the maximum observed concentration of drug.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36, 48, 72, 96, and 120 hours postdose on Day 1
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Moderate Hepatic Impairment | Healthy Control
Number analyzed (Participants) | 10 | 10
ng/mL | 722.6 (293.24) | 802.2 (485.98)
Statistical Analysis 1: Comparison: Moderate Hepatic Impairment vs Healthy Control; An ANOVA model was fitted to the natural logarithmic transformed values of the Cmax. Two-sided 90% CI were calculated for the GLSM ratio of Cmax between hepatic impairment group versus the matched control (normal hepatic function) group; Test type: Other — If the upper bound of the 2-sided 90% CIs of the GLSM ratio for Cmax of filgotinib falls within the [50%, 200%] bound, the null hypothesis that participants with hepatic impairment exhibit Cmax change of at least 2-fold for filgotinib compared with participants with normal liver function will be rejected; GLSM Ratio = 115.98, 90% CI 2-sided [58.75 to 228.98]

6. Primary Outcome: PK Parameter: Cmax of GS-829845
Description: Cmax is defined as the maximum observed concentration of drug. GS-829845 is the primary metabolite of filgotinib.
Time Frame: Predose and 0.5, 1, 2, 3, 4, 5, 6, 8, 12, 18, 24, 36, 48, 72, 96, and 120 hours postdose on Day 1
Population: Participants in the PK Analysis Set were analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Moderate Hepatic Impairment | Healthy Control
Number analyzed (Participants) | 10 | 10
ng/mL | 972.5 (256.09) | 1122.6 (447.45)
Statistical Analysis 1: Comparison: Moderate Hepatic Impairment vs Healthy Control; [analysis description as in outcome 5, analysis 1]; Test type: Other — If the upper bound of the 2-sided 90% CIs of the GLSM ratio for Cmax of GS-829845 falls within the [50%, 200%] bound, the null hypothesis that participants with hepatic impairment exhibit Cmax change of at least 2-fold for GS-829845 compared with participants with normal liver function will be rejected; GLSM Ratio = 102.85, 90% CI 2-sided [60.12 to 175.98]

7. Secondary Outcome: Percentage of Participants Who Experienced Treatment-Emergent Adverse Events
Time Frame: Day 1 up to Day 31
Population: The Safety Analysis Set included all enrolled participants who received at least 1 dose of study drug.
Measure: Number; unit: percentage of participants
Arm/Group | Moderate Hepatic Impairment | Healthy Control
Number analyzed (Participants) | 10 | 10
percentage of participants | 30.0 | 10.0

8. Secondary Outcome: Percentage of Participants Who Experienced Graded Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were defined as values that increase at least one toxicity grade from baseline. The most severe graded abnormality from all tests was counted for each participant.
Time Frame: Day 1 up to Day 31
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Moderate Hepatic Impairment | Healthy Control
Number analyzed (Participants) | 10 | 10
percentage of participants
  Any Laboratory Abnormality | 90.0 | 70.0
  Grade 3 or 4 Laboratory Abnormalities | 60.0 | 0.0

ADVERSE EVENTS:
Time Frame: Day 1 up to Day 31
Description: The Safety Analysis Set included all enrolled participants who received at least 1 dose of study drug.
Arm/Group | Moderate Hepatic Impairment | Healthy Control
All-Cause Mortality (participants affected / at risk) | 0/10 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10
Other Adverse Events (participants affected / at risk) | 3/10 | 1/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Moderate Hepatic Impairment (N=10) | Healthy Control (N=10)
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 0
Rhinitis (Infections and infestations) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2017-12-19): https://cdn.clinicaltrials.gov/large-docs/78/NCT03417778/Prot_000.pdf
  • Statistical Analysis Plan (2018-12-10): https://cdn.clinicaltrials.gov/large-docs/78/NCT03417778/SAP_001.pdf